CLINICAL TRIAL: NCT00841971
Title: Anidulafungin Versus Fluconazole for the Prevention of Invasive Fungal Infections in High-risk Liver Transplant Recipients: a Randomized, Double-blind Trial
Brief Title: Anidulafungin Versus Fluconazole for the Prevention of Fungal Infections in Liver Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Nina Singh, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO08110001
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Mycoses; Fungemia; Central Nervous System Fungal Infections; Lung Diseases, Fungal
MeSH Terms: conditions — Mycoses; Fungemia; Central Nervous System Fungal Infections; Lung Diseases, Fungal | interventions — Anidulafungin; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anidulafungin (Experimental): anti-fungal agent
  Interventions: Drug: Anidulafungin
- Fluconazole (Active Comparator): anti-fungal agent
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Anidulafungin — 200 mg IV loading dose followed by 100 mg qd for 21 days
  Other Names: Eraxis
  Arms: anidulafungin
Drug: Fluconazole — 400 mg IV for 21 days
  Other Names: DIFLUCAN
  Arms: Fluconazole

SUMMARY:
The purpose of this study is to compare the efficacy of anidulafungin versus fluconazole for the prevention of fungal diseases in liver transplant recipients

DETAILED DESCRIPTION:
A number of well characterized risk factors have been shown to portend a high risk of opportunistic mycoses after liver transplantation.

Retransplantation and renal failure are amongst the most significant risk factors for invasive fungal infections in these patients.

Most Invasive fungal infections in these high-risk patients occur within the first month posttransplant.

Studies utilizing universal prophylaxis have primarily employed fluconazole. A recent meta-analysis of prophylactic trials documented a beneficial effect on morbidity and attributable mortality, but an emergence of infections due to non-albicans Candida spp. in patients receiving prophylaxis.

The availability of echinocandins has led to an expanded armamentarium of antifungal drugs with a potentially promising role as agents for targeted prophylaxis for invasive fungal infections in high-risk liver transplant recipients. Anidulafungin is unique amongst echinocandins in that it is eliminated from the body almost exclusively through biotransformation by slow non-enzymatic degradation in the blood, without hepatic metabolism or renal elimination. Anidulafungin has demonstrated good safety profile. We hypothesize that anidulafungin will be more effective and a better tolerated antifungal prophylactic agent in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant recipient at increased risk for infection increased risk include any of the following:
* retransplantation
* renal replacement therapy (dialysis),
* post transplant abdominal surgery (within 21days)
* receipt of corticosteroids for greater than 14 days within the 4 weeks -preceding transplant
* ICU care for greater than 48 hours at the time of transplantation
* colonization with Candida sps within 4 weeks of transplantation
* requirement of 15 units or greater of packed red cell transfusions
* Intraoperative time exceeding 6 hours

Exclusion Criteria:

* Hypersensitivity to azole or echinocandin antifungal agents
* receipt of systemic antifungal therapy within 4 weeks prior to transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2013-07 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Singh, MD, Principal Investigator — University of Pittaburgh, VA Pittsburgh Health Systems
Locations (6):
- United States (6):
  - UCLA Medical Cente, Los Angeles, California
  - University of Miami, Miami, Florida
  - University of Michigan, Ann Arbor, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin

REFERENCES:
- [Result] Winston DJ, Limaye AP, Pelletier S, Safdar N, Morris MI, Meneses K, Busuttil RW, Singh N. Randomized, double-blind trial of anidulafungin versus fluconazole for prophylaxis of invasive fungal infections in high-risk liver transplant recipients. Am J Transplant. 2014 Dec;14(12):2758-64. doi: 10.1111/ajt.12963. Epub 2014 Nov 6. PMID 25376267
- [Derived] Singh N, Winston DJ, Limaye AP, Pelletier S, Safdar N, Morris MI, Meneses K, Busuttil RW, Wagener MM, Wheat LJ. Performance Characteristics of Galactomannan and beta-d-Glucan in High-Risk Liver Transplant Recipients. Transplantation. 2015 Dec;99(12):2543-50. doi: 10.1097/TP.0000000000000763. PMID 26050015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anidulafungin | Fluconazole
Started | 100 | 100
Completed | 98 | 99
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anidulafungin | Fluconazole | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 89 | 178
  >=65 years | 11 | 11 | 22
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [52 to 62] | 58 [51 to 62] | 58 [52 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 28 | 61
  Male | 67 | 72 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 38 | 65
  Not Hispanic or Latino | 73 | 62 | 135
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Fungal Infection
Time Frame: 90 days post enrollment
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 98 | 99
participants | 5 | 8

2. Secondary Outcome: Need for Additional Antifungal Therapy
Time Frame: 90 days post enrollment
Measure: Number; unit: participants
Arm/Group | Anidulafungin | Fluconazole
Number analyzed (Participants) | 98 | 99
participants | 11 | 11

ADVERSE EVENTS:
Arm/Group | Anidulafungin | Fluconazole
Serious Adverse Events (participants affected / at risk) | 1/98 | 0/99
Other Adverse Events (participants affected / at risk) | 11/98 | 11/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anidulafungin (N=98) | Fluconazole (N=99)
Prolonged QT interval (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anidulafungin (N=98) | Fluconazole (N=99)
deaths (General disorders) | 11 (11) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No